CLINICAL TRIAL: NCT01861730
Title: Phase 1/II, Safety and Immunogenicity Study of a Recombinant Protein Tuberculosis Vaccine (AERAS-404) in BCG-Primed Infants
Brief Title: Phase 1/II, Safety and Immunogenicity Study of AERAS-404 in BCG-Primed Infants
Acronym: C-015-404
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Aeras (Other)
Collaborators: Statens Serum Institut (Other); Sanofi Pasteur, a Sanofi Company (Industry); National Institute of Allergy and Infectious Diseases (NIAID) (NIH); International Maternal Pediatric Adolescent AIDS Clinical Trials Group (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: C-015-404/ IMPAACT P1113; U01AI068632 (NIH); C-015-404 (Other: Aeras)
Record Dates: First submitted 2013-05-21; First posted 2013-05-24 (Estimated); Last update posted 2018-04-09 (Actual); Status verified 2018-04

CONDITIONS: Tuberculosis
Keywords: BCG Vaccinated; HIV Negative
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (7):
- Cohort 1 Aeras404 (5ug H4/100nmol IC31) or Placebo (Experimental): 1 Dose; Subject ≥ 168 to ≤ 196 days of age
  Interventions: Biological: AERAS-404; Biological: Placebo
- Cohort 2 AERAS-404 (5ug H4/500nmol IC31) or Placebo (Experimental): 1 Dose; Subject ≥ 168 to ≤ 196 days of age
  Interventions: Biological: AERAS-404; Biological: Placebo
- Cohort 3A AERAS-404 (5ug H4/500nmol IC31) or Placebo (Experimental): 2 Doses; Subject ≥ 168 to ≤ 189 days of age
  Interventions: Biological: AERAS-404; Biological: Placebo
- Cohort 3B AERAS-404 (15ug H4/500nmol IC31) or Placebo (Experimental): 2 Doses; Subject ≥ 168 to ≤ 189 days of age
  Interventions: Biological: AERAS-404; Biological: Placebo
- Cohort 4 AERAS-404 (15ug H4/500nmol IC31) or Placebo (Experimental): 3 Doses; Subject ≥ 84 to ≤ 98 days of age
  Interventions: Biological: AERAS-404; Biological: Placebo
- Cohort 5 AERAS-404 (50ug H4/500nmol IC31) or Placebo (Experimental): 3 Doses; Subject ≥ 84 to ≤ 98 days of age
  Interventions: Biological: AERAS-404; Biological: Placebo
- Cohort 6 AERAS-404 (dose level pending) or Placebo (Experimental): 3 Doses; Subject ≥ 64 to ≤ 83 days of age
  Interventions: Biological: AERAS-404; Biological: Placebo

INTERVENTIONS:
Biological: AERAS-404 — AERAS-404 has two components: the H4 antigen and the IC31 adjuvant. The reconstitution of the vaccine components, H4 antigen (manufactured at SP) and IC31 adjuvant (supplied by SSI), will take place at the clinical research site (CRS) prior to injection.
  Other Names: H4
Biological: Placebo — Tris buffered saline (10mM Tris, pH 7.4, 150nm sodium chloride).
  Other Names: Tris buffered saline

SUMMARY:
Phase I/II, randomized, double-blind, placebo-controlled, safety, immunogenicity and dose-range finding study of AERAS-404 Tuberculosis (TB) vaccine administered intramuscularly in Bacille Calmette-Guerin (BCG) primed infants.

DETAILED DESCRIPTION:
This is a Phase I/II, randomized, double-blind, placebo-controlled, safety, immunogenicity and dose-range finding study in HIV-uninfected, HIV-unexposed, BCG-primed infants. The study vaccine AERAS-404 or placebo will be administered without concomitant EPI vaccines (Cohorts 1 to 5, N = 159 subjects) and with concomitant EPI vaccines (Cohort 6, N = 70 subjects). Study vaccine or placebo will be administered as a single dose (injection) at Study Day 0 ( ≥168 to ≤ 196 days of age, Cohorts 1 and 2), a 2-dose schedule at Study Day 0 (≥ 168 to ≤ 189 days of age) and Study Day 28 (Cohorts 3A and 3B) or a 3-dose schedule at Study Day 0 (≥ 84 to ≤ 98 days of age), Study Day 42 and Study Day 98 (Cohorts 4 and 5). Subjects in Cohort 6 will receive the study vaccine or placebo at Study Day 0 (≥ 64 to ≤ 83 days of age), Study Day 28 (≥ 91 to ≤ 105 days of age), and Study Day 210 (≥ 273 to ≤ 287 days of age). A cohort will enroll once safety in the previous cohort has been established. AERAS-404 is an investigational vaccine manufactured by Sanofi Pasteur (SP) and Statens Serum Institute (SSI).

ELIGIBILITY:
INCLUSION CRITERIA

1. Age at time of entry:

   Cohorts 1 to 6
   * Cohorts 1 and 2: ≥ 168 to ≤ 196 days
   * Cohorts 3A and 3B: ≥ 168 to ≤ 189 days
   * Cohorts 4 and 5: ≥ 84 to ≤ 98 days (≥ 2 weeks after receipt of EPI vaccine doses at 10 weeks of age)
   * Cohort 6 - coincident with EPI vaccine doses at 10 weeks of age (≥ 64 to ≤ 83 days of age)
2. Source documentation of birth weight ≥ 2.5 kg.
3. Documented BCG vaccination within 72 hours of birth.
4. Documented receipt of all age-appropriate EPI vaccines, except Rotavirus, for Cohorts 4 to 6 (see Appendix II).
5. Source documentation of a negative HIV status in the mother, from any time during pregnancy with this child through randomization.
6. Documentation of infant HIV negative exposure or infection status with negative HIV ELISA and HIV DNA PCR tests.
7. Parent or legal guardian able and willing to provide signed informed consent.
8. Participant/parent/legal guardian able to attend all scheduled visits and to comply with all trial procedures.

EXCLUSION CRITERIA

1. History of TB exposure in household or non-household contact.
2. History/Evidence of TB disease or infection.
3. Quantiferon positive.
4. Prior TST test.
5. Any one of Anemia, Neutropenia, Thrombocytopenia, SGPT (ALT), SGOT (AST) or Creatinine ≥ Grade 2
6. Receipt of a live vaccine within 28 days prior to randomization.
7. Receipt or planned receipt of any investigational vaccine.
8. Known or suspected congenital immunodeficiency.
9. Receipt of immunosuppressive therapy or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks within the past 3 months).
10. Known or suspected autoimmune disease
11. Hypersensitivity to any of the vaccine components, or history of a life-threatening reaction to a vaccine containing any of the same substances as the vaccine used in the trial.
12. Participation in another clinical trial for an investigational product (IP).
13. Bleeding disorder or receipt of anticoagulants in the 3 weeks preceding randomization, contraindicating IM vaccination.
14. Chronic illness that, in the opinion of the investigator, is at a stage where it might interfere with trial conduct or completion.
15. Febrile illness (temperature ≥ 100.4°F [≥ 38.0°C]) within 24 hours prior to randomization.

    Note: A subject may enroll after recovery from febrile illness if the subject is still within the age window.
16. Systemic antibiotic use within 48 hours prior to randomization.

Ages: 64 Days to 196 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 243 (Actual)
Dates: Start 2013-07-01 (Actual); Primary Completion 2017-12-22 (Actual); Study Completion 2017-12-22 (Actual)

PRIMARY OUTCOMES:
Investigate the safety of AERAS-404 in HIV-uninfected, HIV-unexposed, BCG-primed infants. | Subjects will be followed for up to 1 year and 4 months.
  Adverse Events and Serious Adverse Events (SAE) will be collected on subjects throughout their participation in the study. Solicited adverse events are captured 28 days post each vaccination. Evaluation of the safety profile of AERAS-404 will be performed using data from all subjects who received at least one dose and has 7 days of safety data, and will be summarized by cohort and treatment group. The number (percentage) of subjects with any adverse event (including solicited, unsolicited, and serious adverse events) will be summarized by Medical Dictionary for Regulatory Activities (MedDRA) system organ class and Preferred Term. Additional summaries will present the number (percentage) of subjects with any adverse events by severity and by relationship to study vaccine; parameters evaluable by the Aeras 404 Pediatric Toxicity Table provided in the protocol, will be summarized by severity corresponding to Toxicity Grade, as appropriate.

SECONDARY OUTCOMES:
Investigate the safety of a 3-dose AERAS-404 regimen in HIV-uninfected, HIV-unexposed, BCG-primed infants | Subjects will be followed for up to 1 year and 4 months.
  The number and percentage of subjects who are enrolled into the three-dose regimen (Cohorts 4-6) with solicited and unsolicited AEs (including serious adverse events [SAEs], local and systemic reactions, and clinical laboratory values or vital sign values recorded as newly abnormal following study vaccination) recorded post-vaccination will be summarized to address the secondary safety objective of the study. Subjects in Cohorts 4 and 5 will be followed for : 1 year and 3 months, Cohort 6: 1 year 4 months and Solicited adverse events are captured 28 days post each vaccination.

OTHER OUTCOMES:
Assess the immunogenicity of a 3-dose AERAS-404 regimen in HIV-uninfected, HIV-unexposed, BCG-primed infants. | Subjects will be followed for up to 1 year and 4 months.
  T-cell response, as measured by Intracellular Cytokine Staining (ICS) following stimulation with peptide pools spanning the vaccine antigens, will be used to assess immunogenicity.
Select an appropriate dose regimen for AERAS-404 in HIV-uninfected, HIV-unexposed, BCG-primed infants. | After all subjects in Cohorts 4 and 5 have completed Study Day 126, the safety and immunogenicity data from these Cohorts will be evaluated. The data will inform the decision on the study vaccine dose for Cohort 6.
  Safety and immunogenicity analyses will be reviewed for the selection of the appropriate dose regimen
Explore interactions between AERAS-404 and EPI vaccines. | Antibody concentration blood samples taken when subjects reach 12 months of age for all Cohorts and in addition, 28 post second study vaccine dose (Study Day 56) for subjects in Cohort 6 only.
  Antibody concentration levels at 12 months of age for all Cohorts, and in addition at 28 days post second study vaccine dose (Study Day 56) for Cohort 6 will be presented. Summaries will include antibody titers to Tetanus toxoid vaccine (tetanus; given at 6, 10, 14 weeks of age), and Haemophilus influenza B conjugate vaccine (given at 6, 10, 14 weeks of age). Responses to other EPI vaccines may also be assessed.
Assess the immunogenicity of a 2-dose AERAS-404 regimen in HIV-uninfected, HIV-unexposed, BCG-primed infants. | Subjects will have Immunology samples taken at multiple time points for up to 1 year and 4 months.

CONTACTS AND LOCATIONS:
Overall Officials: Ann Ginsberg, MD, PhD, Study Director — Aeras; Avy Violari, MD, Principal Investigator — Perinatal HIV Research Unit
Locations (4):
- South Africa (4):
  - PHRU, Chris Hani Baragwanath Hospital, Johannesburg, Guateng
  - Shandukani Research, Johannesburg, Hillbrow
  - KID-CRU, Tygerberg Hospital, Cape Town, Tygerberg
  - South African TB Vaccine Initiative (SATVI), Worcester